CLINICAL TRIAL: NCT06343623
Title: Superiorly Based Pharyngeal Flap Versus Myomucosal Resection and Direct Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, professor of plastic surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fac.med.2018.15
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Velopharyngeal Insufficiency
MeSH Terms: conditions — Velopharyngeal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superiorly based flap (Active Comparator): superiorly bases pharyngeal flap
  Interventions: Procedure: superiorly based flap
- myomucosal resection and direct closure (Experimental): myomucosal resection and direct closure
  Interventions: Procedure: myomucosal resection and direct closure

INTERVENTIONS:
Procedure: myomucosal resection and direct closure — myomucosal resection and direct closure
  Arms: myomucosal resection and direct closure
Procedure: superiorly based flap — superiorly based pharyngeal flap
  Arms: superiorly based flap

SUMMARY:
Patients were classified into two groups. Group (A) patients included fifty patients had velopharyngeal insufficiency and were surgically corrected by the superiorly based pharyngeal flap. Group (B) patients included fifty patients had velopharyngeal insufficiency and were surgically corrected with myomucosal resection and direct closure of the posterior pharyngeal wall

DETAILED DESCRIPTION:
Patients were classified into two groups. Group (A) patients included fifty patients had velopharyngeal insufficiency and were surgically corrected by the superiorly based pharyngeal flap. Group (B) patients included fifty patients had velopharyngeal insufficiency and were surgically corrected with myomucosal resection and direct closure of the posterior pharyngeal wall

ELIGIBILITY:
Inclusion Criteria:

* - Patients have velopharyngeal insufficiency.
* Age range 4-10 years

Exclusion Criteria:

* - Syndromic patients.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
Improvement in the speech outcome | 4 years
  Improvement in the speech outcome using auditory perception assessment and videonasoendoscopy

SECONDARY OUTCOMES:
obstructive sleep apnea | 3 years
  obstructive sleep apnea using respiratory function test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt